CLINICAL TRIAL: NCT01996449
Title: The Role of Aldosterone on Augmented Exercise Pressor Reflex in Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R01HL113738 (NIH)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Hypertension; blood pressure; Aldosterone; Eplerenone; Amlodipine; Primary aldosteronism; Exercise pressor reflex; handgrip exercise; passive arm cycling; active arm cycling
MeSH Terms: conditions — Hypertension; Hyperaldosteronism | interventions — Eplerenone; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial treatment with Amlodipine (Active Comparator): The subject will be started on Amlodipine 2.5-10 mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. The subject will be started on Eplerenone 50 - 200 mg daily, which he or she will continue for a period of 8 weeks. Following the 8 week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Interventions: Drug: Eplerenone; Drug: Amlodipine; Procedure: Microneurography; Procedure: Rhythmic handgrip exercise; Procedure: Sustained hand grip; Procedure: Forearm blood flow; Procedure: Arm cycling exercise; Procedure: Cold Pressor test
- Initial treatment with Eplerenone (Active Comparator): The subject will be started on Eplerenone 50 - 200 mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. The subject will be started on Amlodipine 2.5-10 mg daily, which he or she will continue for a period of 8 weeks. Following the 8 week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Interventions: Drug: Eplerenone; Drug: Amlodipine; Procedure: Microneurography; Procedure: Rhythmic handgrip exercise; Procedure: Sustained hand grip; Procedure: Forearm blood flow; Procedure: Arm cycling exercise; Procedure: Cold Pressor test

INTERVENTIONS:
Drug: Eplerenone — The subject will be started on Eplerenone (Inspra) 50-200mg daily, which he or she will continue for a period of 8 weeks. Following the 8-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued
  Other Names: Inspra
Drug: Amlodipine — The subject will be started on Amlodipine (Norvasc) 2.5 -10mg daily, which he or she will continue for a period of 8 weeks. Following the 8-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Other Names: Norvasc
Procedure: Microneurography — Investigators will measure sympathetic nerve activity from the peroneal nerve by inserting a tiny needle directly into the nerve in the leg. Investigators will localize the nerve by electrical stimulation over the skin using a blunt probe. With this stimulation, subject will notice either involuntary twitching or a tingling sensation, which may be annoying but not painful. Investigators will then introduce a tiny, sterile wire needle (an electrode) through the skin at the same location. When the tip of the needle enters the nerve, subjects may again notice involuntary muscle twitches or tingling in the leg. Investigators will then turn the electrical stimulator off and make minor adjustments in the position of the needle until investigators begin to record the nerve signals. The recording needle will remain in position throughout the study.
  Other Names: Assessment of sympathetic nerve activity (SNA)
Procedure: Rhythmic handgrip exercise — Subjects will perform a rhythmic handgrip exercise at 30% or 45% of maximal voluntary contraction for 3 minutes. Investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure, and sympathetic nerve activity (SNA) at baseline and following this handgrip exercise
Procedure: Sustained hand grip — Subjects will perform a sustained handgrip exercise at 30% of maximal voluntary contraction for 3 minutes. Investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure, and sympathetic nerve activity (SNA) at baseline and following this handgrip exercise.
Procedure: Forearm blood flow — Using high-resolution ultrasound, investigators will measure skeletal muscle blood flow in the forearm at rest, following sustained handgrip exercise
Procedure: Arm cycling exercise — Subjects will perform a cycling arm exercise with a stationary cycling device. Investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure, and sympathetic nerve activity (SNA) at baseline and following this exercise.
Procedure: Cold Pressor test — Subjects will place hand in cold water with ice for 3 minutes. Investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure, and sympathetic nerve activity (SNA) at baseline, during and 2 minutes after the test.

SUMMARY:
Hypertensive patients often show an exaggerated rise in blood pressure during exercise through overactivity of the exercise pressor reflex. An increasing body of evidence suggests a role for aldosterone in augmenting the exercise pressor reflex in hypertensive humans. We hypothesize that this effect of aldosterone is mediated by its direct action on the central nervous system and that administration of mineralocorticoid receptor antagonists constitute an effective treatment for EPR overactivity in hypertension, independent of reductions in resting BP.

DETAILED DESCRIPTION:
Hypertensive patients are known to display exaggerated rise in blood pressure (BP) during exercise but the underlying mechanisms are poorly understood.

Traditionally, muscle afferents were dichotomized as metaboreceptors, which are activated slowly and only during intense or ischemic muscle contraction, or mechanoreceptors, which respond quickly to even mild deformation of their receptive fields. The increase in sympathetic nerve activity and BP caused by activation of these receptors, known as exercise pressor reflex, is normally buffered by activation arterial baroreceptors, which are reset to operate at higher BP range but at the same level of sensitivity. Mechanisms responsible for overactive exercise pressor reflex in hypertension remain unknown, but an increasing body of evidence suggested a role for aldosterone in regulating resting central sympathetic outflow in both hypertensive rats and humans.

Experiments will be performed on 3 groups of subjects 1) stage I (140-159/90-99 mmHg) subjects with essential hypertension, 2) stage I hypertensive subjects with Primary Aldosteronism (PA), and 3) normotensive controls. All participants will attend a baseline study visit, which will include a physical examination, a medical history review, vital sign measurements, and blood and urine collection. Small electrodes will be used to measure muscle nerve activity while the subjects perform a series of exercises that include passive arm cycling, active arm cycling, rhythmic hand grip, sustained hand grip and cold pressor test. Muscle blood flow will be measured before and after hand grip exercises.

A subgroup of subjects with essential hypertension and PA will be assigned to receive Eplerenone or Amlodipine on a randomized, double-blinded design. Participants will attend two weeks visits over a period of 16 weeks. Study visits include measurement of vital signs and blood samples collection. After completing 8 weeks on each medication, muscle nerve activity will be measured while performing the same exercises described in the baseline study visit.

ELIGIBILITY:
Inclusion Criteria:

* Experiments will be performed on 3 groups of nondiabetic human subjects:
* 1) stage I (140-159/90-99 mmHg) subjects with essential hypertension.
* 2) stage I hypertensive subjects with primary aldosteronism
* 3) normotensive controls.

Exclusion Criteria:

* 1) Any evidence of cardiopulmonary disease, left ventricular hypertrophy or systolic dysfunction by echocardiography.
* 2) Blood pressure averaging ≥160/100 mmHg
* 3) Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m2
* 4) Diabetes mellitus or other systemic illness
* 5) Pregnancy
* 6) Hypersensitivity to nitroprusside, phenylephrine, amlodipine or eplerenone
* 7) Any history of substance abuse or current cigarette use
* 8) Any history of psychiatric illness
* 9) History of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Fagard R, Staessen J, Amery A. Maximal aerobic power in essential hypertension. J Hypertens. 1988 Nov;6(11):859-65. doi: 10.1097/00004872-198811000-00003. PMID 3235835
- [Background] Olsen MH, Wachtell K, Hermann KL, Bella JN, Andersen UB, Dige-Petersen H, Rokkedal J, Ibsen H. Maximal exercise capacity is related to cardiovascular structure in patients with longstanding hypertension. A LIFE substudy. Losartan Intervention For Endpoint-Reduction in Hypertension. Am J Hypertens. 2001 Dec;14(12):1205-10. doi: 10.1016/s0895-7061(01)02223-3. PMID 11775128
- [Background] Filipovsky J, Ducimetiere P, Safar ME. Prognostic significance of exercise blood pressure and heart rate in middle-aged men. Hypertension. 1992 Sep;20(3):333-9. doi: 10.1161/01.hyp.20.3.333. PMID 1387630
- [Background] Cleroux J, Beaulieu M, Kouame N, Lacourciere Y. Comparative effects of quinapril, atenolol, and verapamil on blood pressure and forearm hemodynamics during handgrip exercise. Am J Hypertens. 1994 Jun;7(6):566-70. doi: 10.1093/ajh/7.6.566. PMID 7917158
- [Background] Vongpatanasin W, Wang Z, Arbique D, Arbique G, Adams-Huet B, Mitchell JH, Victor RG, Thomas GD. Functional sympatholysis is impaired in hypertensive humans. J Physiol. 2011 Mar 1;589(Pt 5):1209-20. doi: 10.1113/jphysiol.2010.203026. Epub 2011 Jan 4. PMID 21224235
- [Background] Grassi G, Spaziani D, Seravalle G, Bertinieri G, Dell'Oro R, Cuspidi C, Mancia G. Effects of amlodipine on sympathetic nerve traffic and baroreflex control of circulation in heart failure. Hypertension. 1999 Feb;33(2):671-5. doi: 10.1161/01.hyp.33.2.671. PMID 10024325
- [Background] Funder JW, Carey RM, Fardella C, Gomez-Sanchez CE, Mantero F, Stowasser M, Young WF Jr, Montori VM; Endocrine Society. Case detection, diagnosis, and treatment of patients with primary aldosteronism: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2008 Sep;93(9):3266-81. doi: 10.1210/jc.2008-0104. Epub 2008 Jun 13. PMID 18552288

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlodipine Then Eplerenone: The subject will be started on Amlodipine 2.5-10 mg daily, which he or she will continue for a period of 8 weeks. After completion of the study procedures, the medication will be discontinued. The subject will be started on Eplerenone 50 - 200 mg daily, which he or she will continue for a period of 8 weeks.
- Eplerenone Then Amlodipine: The subject will be started on Eplerenone 50 - 200 mg daily, which he or she will continue for a period of 8 weeks. After completion of the study procedures, the medication will be discontinued. The subject will be started on Amlodipine 2.5-10 mg daily, which he or she will continue for a period of 8 weeks.
Period: Period 1: First Drug
Arm/Group | Amlodipine Then Eplerenone | Eplerenone Then Amlodipine
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0
Period: Period 2: Second Drug
Arm/Group | Amlodipine Then Eplerenone | Eplerenone Then Amlodipine
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine Then Eplerenone | Eplerenone Then Amlodipine | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9) | 50 (8) | 51 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Muscle Sympathetic Nerve Activity at Rest
Description: measurement of sympathetic nerve activity by microneurography (intraneural microelectrodes)
Time Frame: 8 weeks post treatment initiation
Measure: Mean (Standard Deviation); unit: bursts/minute
Groups:
- Amlodipine: Analysis independent of sequence. Amlodipine dosage (2.5 -10mg once daily) was titrated every 2 weeks to target BP of < 140/90 mmHg
- Eplerenone: Analysis independent of sequence. Eplerenone dosage (50-200 mg once daily) was titrated every 2 weeks to target BP of < 140/90 mmHg.
Arm/Group | Amlodipine | Eplerenone
Number analyzed (Participants) | 14 | 14
bursts/minute | 41 (11.7) | 43.8 (13)

2. Secondary Outcome: Muscle Sympathetic Nerve Activity During Exercise
Description: measurement of sympathetic nerve activity by microneurography (intraneural microelectrodes) during arm cycling exercise
Time Frame: 8 weeks post treatment initiation
Measure: Mean (Standard Deviation); unit: bursts/minute
Groups:
- Amlodipine; Eplerenone: analysis independent of sequence
Arm/Group | Amlodipine | Eplerenone
Number analyzed (Participants) | 14 | 14
bursts/minute | 47 (16) | 51 (18)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Eplerenone: Analysis independent of sequence. Eplerenone dosage (50 -200mg once daily) was titrated every 2 weeks to target BP of < 140/90 mmHg
Arm/Group | Amlodipine | Eplerenone
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT01996449/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT01996449/ICF_001.pdf